CLINICAL TRIAL: NCT05836987
Title: REACT-AF: Rhythm Evaluation for AntiCoagulaTion With Continuous Monitoring of Atrial Fibrillation
Brief Title: The Rhythm Evaluation for AntiCoagulaTion With Continuous Monitoring of Atrial Fibrillation
Acronym: REACT-AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00354588; 1U24HL165066-01 (NIH)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Anticoagulation; AF-sensing Smart Watch; Ischemic Stroke; Systemic Embolism
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants randomized (1:1) to the experimental arm (AFSW-guided DOAC) will only take DOAC for 30 consecutive days following a qualifying AF episode (i.e., greater than 1 hour) detected by the participants AFSW if no further AF is detected. Participants randomized to the standard of care arm will remain on continuous DOAC throughout the study.
Who Masked: Outcomes Assessor
Masking Description: Adjudication of safety events will be performed by a Clinical Endpoint Committee made up of blinded assessors. The Data Coordinating Center (DCC) blinded statistician(s) will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AFSW Guided DOAC (Experimental): All participants randomized to the experimental arm will be provided with an AFSW that will be linked to the participants Apple watch and the secure REACT-AF app within the Eureka cloud. The AFSW will intermittently and passively assess for rhythm irregularities consistent with AF and notify the wearer and coordinating center if a threshold AF event has occurred.
  Interventions: Device: AFSW Guided DOAC
- Continuous DOAC therapy (Active Comparator): All participants randomized to the control arm will remain on previously prescribed FDA-approved DOAC regimen as indicated by current practice standards. These participants will continuously take DOAC through the course of the study as prescribed by the participants primary physician unless otherwise contraindicated. Participants in the control arm will also use the REACT-AF mobile app within the Eureka platform via Apple watch for study follow-up activities, but the participants will not receive an AFSW and any personally owned Apple Watch will not be loaded with the customized REACT-AF detection algorithm nor participant notification apps.
  Interventions: Drug: Continuous DOAC therapy

INTERVENTIONS:
Device: AFSW Guided DOAC — The AFSW will intermittently and passively assess for rhythm irregularities consistent with AF and notify the wearer and coordinating center if a threshold AF event has occurred.
  Other Names: Apple Watch
  Arms: AFSW Guided DOAC
Drug: Continuous DOAC therapy — DOACs will be prescribed to patients according to the treating healthcare provider(s) according to labeling instructions.
  Other Names: Oral Anticoagulation therapy
  Arms: Continuous DOAC therapy

SUMMARY:
REACT-AF is a multicenter prospective, randomized, open-label, blinded endpoint (PROBE design), controlled trial comparing the current Standard Of Care (SOC) of continuous Direct Oral Anticoagulation (DOAC) use versus time-delimited (1 month) DOAC guided by an AF-sensing Smart Watch (AFSW) in participants with a history of paroxysmal or persistent Atrial Fibrillation (AF) and low-to-moderate stroke risk.

DETAILED DESCRIPTION:
REACT-AF is a prospective, unblinded, randomized (1:1 allocation), multi-center, investigational clinical trial of men and women aged 22-85 with a documented history of symptomatic or asymptomatic paroxysmal or persistent (AF) and a moderate risk of stroke measured by CHA2DS2-VASc score 1-4 for men, 2-4 for women (which stands for Congestive heart failure, Hypertension, Age ≥75 (doubled), Diabetes, Stroke (doubled), Vascular disease, age 65 to 74 and sex category (female)). Participants randomized to the experimental arm (on demand DOAC) will take the participants DOAC for 30 consecutive days following a qualifying AF episode (i.e., greater than1 hour) detected by the AFSW. Participants randomized to the standard of care (control) arm will remain on previously prescribed continuous DOAC throughout the study.

A total of 5350 participants will be enrolled across up to 100 study sites targeting two-thirds academic and one-third private practices, with academic practices also enrolling from affiliated community sites. The investigators anticipate evaluating 7643 consented individuals with external monitoring to ensure that a low AF burden population will be randomized. Up to 200 participants may be enrolled at any one site, and participation will last up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. 22-85 years of age.
2. English speaking participants. Spanish-only speakers may be included in the future at select sites appropriately translated.
3. History of non-permanent atrial fibrillation.
4. CHA2DS2-VASC score of 1-4 for men and 2-4 for women without prior stroke or Transient Ischemic Attack (TIA), The CHA2DS2-VASc score is a point-based system used to stratify the risk of stroke in Atrial Fibrillation (AF) patients. The acronym CHA2DS2-VASc stands for congestive heart failure, hypertension, age ≥75 (doubled), diabetes, stroke (doubled), vascular disease, age 65 to 74 and sex category (female). Congestive heart failure defined as: The presence of signs and symptoms of either right (elevated central venous pressure, hepatomegaly, dependent edema) or left ventricular failure (exertional dyspnea, cough, fatigue, orthopnea, paroxysmal nocturnal dyspnea, cardiac enlargement, rales, gallop rhythm, pulmonary venous congestion) or both, confirmed by non-invasive or invasive measurements demonstrating objective evidence of cardiac dysfunction and/or ejection fraction < 40%.
5. The participant is on a DOAC at the time of screening and willing to stay on DOAC for duration of study.
6. Willing and able to comply with the protocol, including:

   * Possession of a smart watch-compatible smart phone (iPhone that supports the latest shipping iOS) with a cellular service plan
   * Be willing to wear the smart watch for the suggested minimum of 14 hours a day
   * Expected to be within cellular service range at least 80% of the time
7. Willing and able to discontinue DOAC
8. The participant is willing and able to provide informed consent.

Exclusion Criteria:

1. Valvular or permanent atrial fibrillation.
2. Current treatment with warfarin and unwilling or unable to take a DOAC.
3. The participant is a woman who is pregnant or nursing.
4. The participant is being treated with chronic aspirin, another anti-platelet agent, or chronic NSAIDS outside of current medical guidelines (e.g., primary stroke prevention in patients with atrial fibrillation, primary prevention of cardiovascular events, pain relief, fever, gout) and is unwilling or unable to discontinue use for the study duration.
5. Existing cardiac rhythm device or indication for a permanent pacemaker, Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy (CRT) device or planned insertable cardiac monitor. Insertable cardiac monitors are permitted unless they are being used to guide anticoagulation treatment.
6. Known or suspected symptomatic or asymptomatic atrial fibrillation lasting ≥ 1 hour/month over the last 3 months.
7. Any documented single AF episode lasting ≥ 1 hour on standard of care or study-provided external cardiac monitor of > 6 days duration performed within 45 days prior to randomization. Shorter monitoring durations may be acceptable for inclusion at the discretion of the site PI based on the totality of monitoring data and approval of the study PI.
8. Ablation for AF within the last 2 months.
9. Prior or anticipated left atrial appendage occlusion or ligation.
10. Mechanical prosthetic valve(s) or severe valve disease.
11. Hypertrophic cardiomyopathy.
12. Participant needs DOAC for reasons other than preventing stroke or arterial embolism resulting from AF (i.e., preventing Deep Vein Thrombosis (DVT) or PE) or needs permanent OAC (i.e., congenital heart defects, prosthetic heart valve).
13. Participants deemed high risk for non-cardioembolic stroke (i.e., significant carotid artery disease defined as stenosis > 75%) based on the investigator's discretion.
14. The participant is enrolled, has participated within the last 30 days, or is planning to participate in a concurrent drug and/or device study during the course of this clinical trial. Co-enrollment in concurrent trials is only allowed with documented pre-approval from the study manager; there is no concern that co-enrollment could confound the results of this trial.
15. The participant has a tattoo, birthmark, or surgical scar over the dorsal wrist area on the ipsilateral side that the AFSW may be worn.
16. The participant has a tremor on their ipsilateral side that the AFSW may be worn.
17. Any concomitant condition that, in the investigator's opinion, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse).
18. Known hypersensitivity or contraindication to direct oral anticoagulants.
19. Documented prior stroke (ischemic or hemorrhagic) or transient ischemic attack.
20. Reversible causes of AF (e.g., cardiac surgery, pulmonary embolism, untreated hyperthyroidism). AF ablation does not constitute reversible AF.
21. > 5% burden of premature atrial or ventricular depolarizations on pre-enrollment cardiac monitoring.
22. History of atrial flutter that has not been treated with ablation (participants in atrial flutter and have been ablated are eligible for enrollment).
23. Stage 4 or 5 chronic kidney disease.
24. Conditions associated with an increased risk of bleeding:

    * Major surgery in the previous month
    * Planned surgery or intervention in the next three months that would require cessation of anticoagulation > 2 weeks.
    * History of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intra- articular bleeding
    * Gastrointestinal hemorrhage within the past year unless the cause has been permanently eliminated (e.g., by surgery)
    * Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days
    * Hemorrhagic disorder or bleeding diathesis
    * Need for anticoagulant treatment for disorders other than AF
    * Uncontrolled hypertension (Systolic Blood Pressure >180 mmHg and/or Diastolic Blood Pressure >100 mmHg)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5350 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess whether AFSW-guided, time-delimited DOAC therapy is non-inferior to continuous DOAC therapy for a composite endpoint that includes: (1) Ischemic stroke; (2) Systemic embolism; (3) All-cause mortality. | At 60 months
  The primary objective (efficacy objective) of the REACT-AF trial is to assess whether AFSW-guided, time-delimited DOAC therapy is non-inferior to continuous DOAC therapy for a composite endpoint that includes: (1) Ischemic stroke; (2) Systemic embolism; and (3) All-cause mortality.
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction; and classified as ischemic, hemorrhagic, or cause unknown based on CT or Magnetic Resonance (MR) scanning or autopsy.
  Systemic embolism is defined as an acute vascular occlusion of the extremities or any organ and must be documented by angiography, surgery, scintigraphy, or autopsy and require hospitalization.
  All-cause mortality will be defined as the underlying disease or injury that initiates the train of events resulting in death.

SECONDARY OUTCOMES:
To assess whether AFSW-guided, time-delimited DOAC therapy significantly reduces major bleeding events compared to continuous DOAC therapy. | At 60 months
  Oral anticoagulation carries a risk of major bleeding, including life-threatening hemorrhage, the intervention is expected to reduce the safety endpoint, major bleeding, by > 35%, and the study is powered for the superiority of the safety endpoint.
  Major bleeding will be defined as requiring hospitalization and by ≥1 of the following International Society on Thrombosis and Haemostasis (ISTH) criteria: (1) Bleeding associated with a reduction in hemoglobin level of at least 2.0 g/dL; (2) Bleeding leading to transfusion of at least two units of blood or packed cells; or (3) Symptomatic bleeding in a critical area or organ such as intraocular, intracranial, intraspinal or intramuscular with compartment syndrome, retroperitoneal bleeding, intra-articular bleeding, or pericardial bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Rod Passman, Principal Investigator — Northwestern University; Dan Hanley, Principal Investigator — Johns Hopkins University
Locations (91):
- United States (91):
  - Banner University, Phoenix, Arizona
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - University of California Los Angeles (UCLA Health), Los Angeles, California
  - UC Davis Health, Sacramento, California
  - Scripps Health, San Diego, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - South Denver Cardiology Associates, P.C., Littleton, Colorado
  - St. Elizabeth's Medical Center, Washington D.C., District of Columbia
  - Medical Faculty Associates George Washington University, Washington D.C., District of Columbia
  - BayCare Health Systems, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami - Leonard S. Miller SOM, Miami, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Cleveland Clinic Florida, Stuart, Florida
  - Baycare Health Systems Clearwater, Winter Haven, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Arrhythmia Consultants and Research Institute, Warner Robins, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Chicago, Illinois
  - Alexian Brothers Health System, Elk Grove Village, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Maine Medical Partners MaineHealth Cardiology, Scarborough, Maine
  - Johns Hopkins Univeristy, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mass General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - BMC - Brighton, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - UMass Chan Medical School, Worcester, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Corewell Health (Former Spectrum Health), Grand Rapids, Michigan
  - Trinity Health Grand Rapids/Mercy Health, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Trinity Health Michigan Heart - Ann Arbor, Ypsilanti, Michigan
  - Essentia Health The Duluth Clinic, Duluth, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University Health Truman Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Advanced Heart and Vascular Institute of Hunterdon, Flemington, New Jersey
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Rutgers, the State University of New Jersey, Piscataway, New Jersey
  - The Valley Hospital, Inc., Ridgewood, New Jersey
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Presbyterian Healthcare Services, Albuquerque, New Mexico
  - University at Buffalo, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - NewYork Presbyterian - Queens, Queens, New York
  - Staten Island University Hospital-Northwell Health, Staten Island, New York
  - Stony Brook University, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - White Plains Hospital, White Plains, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Wooster Community Hospital, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Penn State Health Medical Group Berks Cardiology, Wyomissing, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Health Heart and Vascular, Columbia, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - James River Cardiology, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - St. Joseph Medical Center Tacoma, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin